CLINICAL TRIAL: NCT01446458
Title: Phase I Study of Stereotactic Body Radiation Therapy and 5-Fluorouracil, Oxaliplatin and Irinotecan (FOLFIRINOX) in the Neoadjuvant Therapy of Pancreatic Cancer
Brief Title: Phase I Study of Stereotactic Body Radiation Therapy and FOLFIRINOX in the Neoadjuvant Therapy of Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Natalyn N. Hawk, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00051215; WCI1998-11 (Other: Other)
Record Dates: First submitted 2011-09-26; First posted 2011-10-05 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Cancer of Pancreas; Cancer of the Pancreas; Neoplasms, Pancreatic; Pancreas Cancer; Pancreas Neoplasms
Keywords: Cancer of Pancreas; Cancer of the Pancreas; Neoplasms, Pancreatic; Pancreas Cancer; Pancreas Neoplasms; Entry Term Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5-Fluorouracil, Oxaliplatin, Irinotecan (Experimental): 5-Fluorouracil, Oxaliplatin, Irinotecan are administered as a modified FOLFIRINOX regimen every 15 days. Subjects receive bi-weekly cycles of therapy on the 1st week, the 3rd week, the 5th week and finally the 7th week for a total of 4 cycles. Assessments include history and physical, laboratory tests on a weekly basis throughout the treatment period prior to and including week 8 assessment for stereotactic body radiotherapy (SBRT).
  Interventions: Drug: Modified FOLFIRINOX; Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Drug: Modified FOLFIRINOX — Patients receive modified FOLFIRINOX Chemotherapy for 4 cycles (1 cycle = 15 days). Modified FOLFIRINOX: Oxaliplatin 85 mg/m2 intravenous infusion on day 1; Irinotecan 180 mg/m2 intravenous infusion on day 1; 5-Fluorouracil 2400 mg/m2 continuous intravenous infusion on days 1 to 3; pegylated filgrastim (neulasta) 6 mg subcutaneous injection on day 3.
  Other Names: modifiedFOLFIRINOX
Radiation: Stereotactic Body Radiotherapy (SBRT) — Patients will receive Stereotactic Body Radiotherapy (SBRT) to pancreas tumor 2 weeks following chemotherapy. SBRT is given in 3 daily fractions at designated doses per treatment cohort. Starting dose level-Dose level 1: 10 Gy SBRT to primary tumor volume (PTV) / 2 Gy SBRT to the retroperitoneal margin daily for a total Gy to Gross tumor volume (GTV) of 36 Gy. There are weekly toxicity assessments for 4 weeks. This is a standard 3 + 3 design with 4 dose levels.
  Other Names: SBRT

SUMMARY:
The purpose of this study is to determine whether using FOLFIRINOX chemotherapy and Stereotactic Body Radiation Therapy (SBRT) prior to surgery in patients with pancreatic cancer is safe and well tolerated. This study will obtain preliminary data on the response of the cancer to this therapy by Magnetic Resonance Imaging (MRI) and by studying the cancer after it is resected surgically.

In addition, the investigators will perform biochemical studies on the tumor tissue obtained from your tissue biopsy as well as from the tumor removed by the surgeon in order to measure the effect of treatment with FOLFIRINOX and SBRT on several proteins that may be important in the behavior of pancreatic cancer cells.

The data obtained from this trial will be extremely valuable to help improve the approach to treating pancreatic cancer in the future. If you do not undergo surgery after completion of FOLFIRINOX + SBRT, the investigators will request a second biopsy of the tumor under computer tomography (CT) -guidance in order to measure the effect of treatment on your tumor.

DETAILED DESCRIPTION:
The current standard of care for treating early stage pancreatic cancer involves surgery followed by chemotherapy and / or chemoradiotherapy using conventional fractionated external beam radiation therapy (EBRT). Despite the the incorporation of multi-modality adjuvant therapy following surgery, patients with surgically resected pancreas cancer have a high likelihood of recurrence of their cancer and/ or death from their disease. Patients with more advanced pancreatic cancers experience even worse outcomes in the face of unresectable disease or lower likelihood of achieving a negative margin resection. In these particular group of patients, chemotherapy and radiation given prior to surgery may help select patients who are more likely ultimately to benefit from a pancreaticoduodenectomy and may improve the rate of margin negative resection, factors which may influence their outcome.

Systemic chemotherapy traditionally used in the treatment of pancreatic cancer has included drugs such as gemcitabine or 5-fluorouracil (5-FU). Recently, a multi-agent chemotherapy regimen called FOLFIRINOX has shown significant efficacy in patients with advanced pancreatic cancer with improved tumor responses and improved overall outcomes with a reasonable toxicity profile.

Stereotactic body radiotherapy (SBRT) is a unique radiation technique that allows higher doses of radiation to be delivered to the cancer over a significantly shorter period of time compared to conventional radiation. SBRT's advantages over conventional radiation include: shorter duration of therapy (one to three days versus two to five weeks) as well as the ability to deliver full doses of chemotherapy. In treating patients with pancreatic cancer, SBRT has been tolerated and has been effective when compared historically to conventional radiation. SBRT has been combined with chemotherapy and has also been very well tolerated in patients with pancreatic cancer.

This study will ask whether giving chemotherapy with FOLFIRINOX followed in short sequence by radiation therapy using Stereotactic Body Radiation Therapy (SBRT) is safe and feasible. This study will also begin to ask what is the effect of this approach on the rate of margin negative resection in patients who may subsequently undergo surgery for their pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria: Patients eligible must have:

* Histologic or cytologic diagnosis of pancreatic adenocarcinoma.
* Radiographically resectable or borderline resectable disease as reviewed by an experienced surgical oncologist at Emory.
* Age 21 years or older.
* Not received prior chemotherapy or radiation for pancreatic cancer.
* ECOG performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Adequate bone marrow function: absolute neutrophil count > 1,500/cmm, platelet count > 100,000/cmm.
* Understanding and be informed of the investigational nature of this study and must give written informed consent prior to the receiving of treatment per this protocol.

Exclusion Criteria: Patients who are not eligible have

* Histologies including endocrine tumors or lymphoma of the pancreas.
* A tumor which is less than 3 mm from the duodenum as measured by either CT or MRI.
* History of central nervous system (CNS) metastases.
* Liver dysfunction, including total bilirubin > 1.5 mg/dL; aspartate transaminase (AST) and alanine amino transferase (ALT) > 5 times upper limit of the institutional normal.
* Creatinine ≥ 1.5 mg/dL.
* Albumin ≤ 2.5 g/dL.
* International Normalized Ratio (INR) ≥ 1.5 (in the absence of ongoing treatment with warfarin).
* Breast feeding.
* Serious active infection.
* Serious concurrent systemic disorders incompatible with participating in the study (at the discretion of the investigator).
* An active second primary malignancy (except in situ carcinoma of the cervix, or adequately treated basal cell carcinoma of the skin) within less than one year of enrollment into this study.
* Clinical evidence of distant metastatic disease.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated total dose of stereotactic body radiation to patients with resectable or borderline resectable pancreas cancer following FOLFIRINOX chemotherapy | Four weeks
  A standard 3 + 3 design will be used for evaluating the safety and tolerability of SBRT radiation doses. Any grade 3 liver, gastric, small bowel or spinal cord toxicity or any grade 4 toxicity (hematologic or other non-hematologic except for diarrhea) will be considered a dose limiting toxicity (DLT).
  Each cohort will consist of 3 patients, unless 1 of the patients experiences a DLT in which case the cohort will be expanded to 6 patients. The maximum tolerated dose (MTD) will be defined as the dose level below that which results in a DLT in 2 or more of the 6 patients in a cohort.

SECONDARY OUTCOMES:
Clinical and pathologic objective response rate as measured by MRI (clinical response) and histopathology and rate of complete resection (R0) (pathologic response) | ten weeks
  The overall pathologic (complete + partial) response rate and margin negative resection rate will be estimated using all registered patients and all resected patients (via the Intention to Treat principle for effectiveness assessment).
  The overall objective clinical response rate will involve MRI assessment of pancreas tumors of all registered patients with comparison of baseline (pre-treatment) MRI measurement to post-treatment MRI measurement prior to surgical resection using the Response Evaluation Criteria in Solid Tumors (RECIST). Measurements will involve all registered patients.

CONTACTS AND LOCATIONS:
Overall Officials: Natalyn N. Hawk, MD, PhD, Principal Investigator — Emory University Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia

REFERENCES:
- [Derived] Shaib WL, Hawk N, Cassidy RJ, Chen Z, Zhang C, Brutcher E, Kooby D, Maithel SK, Sarmiento JM, Landry J, El-Rayes BF. A Phase 1 Study of Stereotactic Body Radiation Therapy Dose Escalation for Borderline Resectable Pancreatic Cancer After Modified FOLFIRINOX (NCT01446458). Int J Radiat Oncol Biol Phys. 2016 Oct 1;96(2):296-303. doi: 10.1016/j.ijrobp.2016.05.010. Epub 2016 May 24. PMID 27475674